CLINICAL TRIAL: NCT03420547
Title: Renewing Intimacy and Sexuality (RISE): a Pilot Program to Support Marital Intimacy and Sexual Health of Female Cancer Patients in Singapore
Brief Title: Marital Satisfaction and Sexual Health of Female Cancer Patients in Singapore
Acronym: RISE
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Duke-NUS Graduate Medical School (Other)
Responsible Party: Principal Investigator, Irene Teo, Assistant Professor, Duke-NUS Graduate Medical School
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: Duke-NUS
Record Dates: First submitted 2018-01-16; First posted 2018-02-05 (Actual); Last update posted 2025-02-05 (Actual); Status verified 2025-02

CONDITIONS: Gynecologic Cancer; Breast Cancer
MeSH Terms: conditions — Breast Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Intervention group (Experimental): Group of participants receiving the RISE intervention
  Interventions: Behavioral: RISE
- Standard Care (waitlist) (No Intervention): Group receiving no intervention in first 6 weeks.They will have the option of participating in the RISE program after their second assessment at week 6.

INTERVENTIONS:
Behavioral: RISE — Intervention will consist of 3 sessions over 6 weeks. Each session will last 2 hours and be conducted with a clinical psychologist or medical social worker. The intervention content include psycho-education, communication training between the couple, and exercises to foster intimacy. A therapy manual will be developed to ensure program delivery fidelity. A folder with session summaries will be provided to the participants.The intervention content include psycho-education, communication training between the couple, and exercises to foster intimacy. A therapy manual will be developed to ensure program delivery fidelity. A folder with session summaries will be provided to the participants.
  Arms: Intervention group

SUMMARY:
Disturbances in marital intimacy and sexual health is one of the most underrated and undertreated problems in cancer survivorship. A review on unmet supportive care needs of cancer patients noted one third to more than half of patients reported support for sexual disturbances as an area of unmet need during and after treatment. Patients, whose sense of femininity and body image may be at risk, such as in the case of breast and gynaecologic cancers, may be more susceptible to such intimacy and sexual disturbances. According to a recent study conducted in Singapore, 25% of gynaecologic cancer patients reported dissatisfaction with their bodies and 19% reported feeling less sexually attractive. Unfortunately, there is paucity in formal resources for couples counselling within the oncology setting in Singapore. The current study seeks to investigate a pilot program called Renewing Intimacy and Sexuality (RISE), which consists of 3 sessions with female cancer patients and their spouses, and that combine components of psychosexual education, communication training and skills building. The reach, acceptability, implementation, and preliminary effectiveness of the RISE program will be assessed based on the RE-AIM framework for program planning. The overall aim of the research project is to establish evidence-based programs for cancer survivors to enhance their quality of life.

DETAILED DESCRIPTION:
This is a multi-site, randomized controlled, pilot intervention study. Patients seen in outpatient clinics in the Department of Gynaecologic Oncology at KKH Women and Children's Hospital (KKH) and the breast team within the Division of Medical Oncology at National Cancer Centre (NCC) will be recruited to participate. Patients who meet pre-screen criteria will be invited to complete a self-report screener of marital and sexual well-being. Those who are eligible for the study and indicate interest will be contacted to participate in the RISE program. Study participants will sign an informed consent before being given a pre-treatment assessment and being randomized using an opaque, sealed envelope system to receive either (i) the RISE program or (ii) Standard Care. Those in the Standard Care group will have the option of participating in the RISE program after their second pre-treatment assessment to ensure all participants are given the opportunity to receive the program. Randomization is stratified by cancer (i.e., gynaecologic vs breast) and occur in permuted blocks. At the end of participation in the RISE program, all participants will be given a post-treatment assessment. Spouse of the participants will be invited to participate in the study. Those who agree will complete a pre-treatment survey similar to the patient participant and attend the 3 sessions with the patient, and complete a post-treatment assessment similar to the patient's.

The RISE Intervention consists of 3 sessions which will last 2 hours each and be conducted with a clinical psychologist or medical social worker with experience with couples counseling. The intervention content include psycho-education, communication training between the couple, and exercises to foster intimacy. A therapy manual will be developed to ensure program delivery fidelity. A folder with session summaries will be provided to the participants.

ELIGIBILITY:
Inclusion Criteria:

1. Aged 21 years or old
2. Has a spouse/ romantic partner
3. History of stage I-III gynaecologic or breast cancer
4. At least 4 weeks post completion of active treatment (i.e., surgery, chemotherapy, radiation therapy)
5. Patient meets cut-off for marital distress on the Dyadic Adjustment Scale-4 (defined as overall score of ≤ 12) or sexual distress (defined as endorsing "occasionally" - "always" to the question how often patient felt distress about their sex life in the last 30 days)
6. Speak and read English

Exclusion Criteria:

1. Diagnosis of metastatic (stage IV) cancer
2. Visual, hearing, or cognitive impairment that will interfere with participation

   -

Ages: 21 Years to 100 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes
Enrollment: 41 (Actual)
Dates: Start 2018-11-01 (Actual); Primary Completion 2022-07-31 (Actual); Study Completion 2024-01-01 (Actual)

PRIMARY OUTCOMES:
Assess the reach of the RISE program | Baseline
  Measured by proportion of those who enrol to those who are eligible to participate.
Determine the acceptability of the RISE program | Week 6 for intervention arm; Week 12 for waitlist arm
  Measured by participant rated satisfaction with the program using the Client Satisfaction Questionnaire
Success of implementation of the program. | Week 6 for intervention arm; Week 12 for waitlist arm
  Measured by participant's willingness to pay for the program.
Collect feedback to improve the RISE program | Week 6 for intervention arm; Week 12 for waitlist arm
  Obtained by conducting semi-structured interviews with participants at program completion.

SECONDARY OUTCOMES:
Preliminary data on effectiveness of the program. | Change in scores from Baseline to Week 6 for intervention arm; change in scores from Baseline to Week 12 for Waitlist arm
  Measured by change in relationship well-being using the Dyadic Adjustment Scale-10

CONTACTS AND LOCATIONS:
Overall Officials: Irene Teo, PhD, Principal Investigator — Duke-NUS Graduate Medical School
Locations (2):
- Singapore (2):
  - KK Women's and Children's Hospital, Singapore, Singapore
  - National Cancer Centre, Singapore

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Glasgow RE, McKay HG, Piette JD, Reynolds KD. The RE-AIM framework for evaluating interventions: what can it tell us about approaches to chronic illness management? Patient Educ Couns. 2001 Aug;44(2):119-27. doi: 10.1016/s0738-3991(00)00186-5. PMID 11479052
- [Background] Teo I, Cheung YB, Lim TYK, Namuduri RP, Long V, Tewani K. The relationship between symptom prevalence, body image, and quality of life in Asian gynecologic cancer patients. Psychooncology. 2018 Jan;27(1):69-74. doi: 10.1002/pon.4457. Epub 2017 Jun 16. PMID 28508411
- [Derived] Teo I, Tan YP, Goh A, Pan FT, Tan TJ, Ozdemir S, Cheung YB, Chaudhry I, Razali NS, Tewani KG. The Renewing Intimacy and SExuality Intervention for Female Cancer Survivors: A Feasibility Study. Psychooncology. 2024 Dec;33(12):e70037. doi: 10.1002/pon.70037. PMID 39638564